CLINICAL TRIAL: NCT02780687
Title: LUX-Bladder 1: Phase II Open Label Single Arm Exploratory Trial of Oral Afatinib Monotherapy Following Platinum Failure for Patients With Advanced/Metastatic Urothelial Tract Carcinoma With Genetic Alterations in ERBB Receptors.
Brief Title: Afatinib Monotherapy in Patients With ERBB-deregulated Metastatic Urothelial Tract Carcinoma After Failure of Platinum Based Chemotherapy
Acronym: LUX-Bladder 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.261; 2015-005427-10 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental)
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib

SUMMARY:
The purpose of this trial is to assess the anti-tumour activity and safety of afatinib monotherapy in patients with urothelial tract carcinoma carrying ERBB2 or ERBB3 (Erythroblastic leukaemia viral oncogene homolog of the human epidermal growth factor family of receptors) mutations or ERBB2 amplifications (Cohort A), and EGFR (Epidermal Growth Factor Receptor) amplification positive tumours (Cohort B), progressing despite previous platinum based chemotherapy, and thereby to improve their prognosis.

The antitumour activity of afatinib monotherapy in these patients will be assessed by progression free survival rate at 6 months (PFS6). This will be the primary endpoint of the trial. A key secondary endpoint will also be defined, the objective response rate (ORR).

ELIGIBILITY:
Inclusion criteria:

* Recurrent or metastatic urothelial cancer
* Patients must have failed prior platinum based treatment (adjuvant or 1st line)
* Archival tissue sample available for biomarker testing at pre-screening and tissue banking.
* Patients should complete a pre-screening biomarker analysis and should fulfill the following: for Cohort A tumour should show a ERBB2 (epidermal growth factor family receptor 2) or ERBB3 mutation, or ERBB2 gene amplification; for Cohort B tumour should show EGFR (Epidermal Growth Factor Receptor) amplification.
* Further inclusion criteria apply

Exclusion criteria:

* Prior use of EGFR, ERBB2 or ERBB3 targeted treatment
* Chemotherapy within 4 weeks prior to the start of study treatment. Biological therapy or investigational agents within 4 weeks prior to the start of study treatment or prior to passing 5 half-lives, i.e. systemic clearance, whatever comes first
* Known brain metastases or signs hereof, uncontrolled spinal cord compression or leptomeningeal carcinomatosis
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- France (9):
  - INS Bergonié, Bordeaux
  - CTR Leon Berard, Lyon
  - INS Cancérologie du Gard, Nîmes
  - HOP Saint-Louis, Paris
  - HOP Cochin, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Foch, Suresnes
  - INS Universitaire du Cancer, Toulouse
  - INS Gustave Roussy, Villejuif
- Italy (2):
  - Ospedale San Donato di Arezzo, Arezzo
  - A.O. San Camillo Forlanini, Roma
- Spain (19):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de Elche, Elche
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - CIO Clara Campal, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - CS Parc Taulí, Sabadell
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Derived] Font A, Mellado B, Climent MA, Virizuela JA, Oudard S, Puente J, Castellano D, Gonzalez-Del-Alba A, Pinto A, Morales-Barrera R, Rodriguez-Vida A, Fernandez PL, Teixido C, Jares P, Aldecoa I, Gibson N, Solca F, Mondal S, Lorence RM, Serra J, Real FX. Phase II trial of afatinib in patients with advanced urothelial carcinoma with genetic alterations in ERBB1-3 (LUX-Bladder 1). Br J Cancer. 2024 Feb;130(3):434-441. doi: 10.1038/s41416-023-02513-6. Epub 2023 Dec 15. PMID 38102226
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a Phase II open label single arm exploratory trial of oral afatinib monotherapy following platinum failure for patients with advanced/metastatic urothelial tract carcinoma with genetic alterations in ERBB receptors.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Cohort A: Afatinib monotherapy in patients with urothelial tract carcinoma who progressed after first line of platinum-based chemotherapy and who show mutations in ERBB2 or ERBB3 or amplification in ERBB2 (Erythroblastic leukaemia viral oncogene homolog of the human epidermal growth factor family of receptors). Therapy consists of 40 mg film-coated tablets taken orally once a day continuously. The dose could be reduced to 30 mg or, in a second step, to 20 mg once daily. No dose increase was allowed after a dose reduction.
- Cohort B: Afatinib monotherapy in patients with urothelial tract carcinoma who progressed after first line of platinum-based chemotherapy and who show EGFR (Epidermal Growth Factor Receptor) amplification. Therapy consists of 40 mg film-coated tablets taken orally once a day continuously. The dose could be reduced to 30 mg or, in a second step, to 20 mg once daily. No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 34 | 8
Completed | 0 | 0
Not Completed | 34 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Switched to commercial program (in CTP) | 2 | 0
Not completed — progressive disease | 29 | 6

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all patients who took at least 1 afatinib dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 34 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.3) | 70.0 (6.9) | 67.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 30 | 6 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 8 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Biomarker status [Number; unit: Participants]
  ERBB2 mutation | 8 | 0 | 8
  ERBB3 mutation | 11 | 0 | 11
  ERBB2 amplification | 20 | 0 | 20
  EGFR amplification | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival at Six Months (PFS6) in Cohort A
Description: Progression-free survival at 6 months for Cohort A was defined as the number of patients who were alive and without disease progression at 24-week tumour assessment. Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated. Progression is defined as at least a 20% increase in sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD since the treatment started, together with an absolute increase in the sum of LD of at least 5 millimeter OR The appearance of one or more new lesions.
Time Frame: From start of treatment till assesment at week 24.
Population: The treated set (TS) included all patients who took at least 1 afatinib dose. The aim of the study was to investigate patients with ERBB-deregulated tumours (cohort A), patients with EGFR amplification (cohort B) were therefore not included in the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Participants
  Without progression/death at 24th week | 4

2. Secondary Outcome: Number of Participants With Confirmed Objective Response (ORR) in Cohort A
Description: Confirmed objective response by investigator review for Cohort A was defined as the number of participants with confirmed complete response (CR, disappearance of all target lesions) or confirmed partial response (PR, at least a 30% decrease in sum of longest diameter (LD) of target lesions, reference is baseline sum LD). Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated.
Time Frame: Scans every 8 (±1) weeks from start till end of treatment. Afterwards, if discontinuation was not for progression: every 8 (±1) weeks until month 6, every 12 (±2) weeks thereafter. Until documented disease progression, i.e., up to ~ 20 Months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Participants
  Objective response | 2

3. Secondary Outcome: Progression-free Survival (PFS) in Cohort A
Description: Progression-free survival was defined as the time (months) from the date of the first afatinib administration to the date of disease progression or death (if the patient died without progression). The date of progression for the primary analyses was determined based on investigator assessment. Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to RECIST version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated. Progression is defined as at least a 20% increase in sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD since the treatment started, together with an absolute increase in the sum of LD of at least 5 millimeter OR The appearance of one or more new lesions.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Weeks | 9.8 [7.9 to 16.0]

4. Secondary Outcome: Overall Survival (OS) in Cohort A
Description: Overall survival (OS) defined as the time from start of treatment of afatinib until death from any cause.
Time Frame: From start of treatment of afatinib until death from any cause, i.e. up to approximately 20 Months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Weeks | 30.1 [17.4 to 47.0]

5. Secondary Outcome: Number of Participants With Disease Control (DCR) in Cohort A
Description: Disease control was calculated as the number of participants with complete response (CR, disappearance of all target lesions), partial response (PR, at least a 30% decrease in sum of longest diameter (LD) of target lesions, reference is baseline sum LD), or stable disease (SD, neither sufficient shrinkage to qualify for PR, taking as reference the baseline sum of diameters (SoD), nor sufficient increase to qualify for PD (Progression) taking as reference the smallest SoD since the treatment started). Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Participants
  Yes | 17
  No | 17

6. Secondary Outcome: Duration of Disease Control in Cohort A
Description: For patients with disease control, duration of disease control was defined as the time from afatinib treatment start to disease progression (or death if the patient died before progression).
  Disease control was defined as a having a complete response (CR, disappearance of all target lesions), partial response (PR, at least a 30% decrease in sum of longest diameter (LD) of target lesions, reference is baseline sum LD), or stable disease (SD, neither sufficient shrinkage to qualify for PR, taking as reference the baseline sum of diameters (SoD), nor sufficient increase to qualify for PD taking as reference the smallest SoD since the treatment started). Tumour response was assessed based on local radiological image (CT or MRI) evaluation by the investigators according to RECIST version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Weeks | 22.7 [15.1 to 36.1]

7. Secondary Outcome: Number of Patients With Tumour Shrinkage in Cohort A
Description: Number of patients with tumour shrinkage, tumour shrinkage from baseline was defined by the maximum percentage decrease from baseline in the sum of the longest diameters of target lesions. Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Baseline imaging was to be performed within 28 days before afatinib treatment start, if the patient already had a tumour assessment within this timeframe, this test was not repeated.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 34
Participants
  Patients with Shrinkage | 9

ADVERSE EVENTS:
Time Frame: From the time of first drug administration till the end of treatment + 30 days (REP), up to approximately 20 Months.
Description: The treated set (TS) included all patients who took at least 1 afatinib dose.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 26/34 | 7/8
Serious Adverse Events (participants affected / at risk) | 15/34 | 6/8
Other Adverse Events (participants affected / at risk) | 34/34 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=34) | Cohort B (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=34) | Cohort B (N=8)
Anaemia (Blood and lymphatic system disorders) | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 10 | 1
Diarrhoea (Gastrointestinal disorders) | 23 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 1
Stomatitis (Gastrointestinal disorders) | 9 | 2
Vomiting (Gastrointestinal disorders) | 7 | 1
Asthenia (General disorders) | 19 | 3
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 10 | 3
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 7 | 1
Xerosis (General disorders) | 3 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 2 | 0
Skin candida (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Leukocyturia (Renal and urinary disorders) | 2 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 11 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 4 | 1
Hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Duration of confirmed objective response was not analysed because only 2 patients showed a confirmed objective response. Instead, duration of disease control was analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT02780687/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT02780687/SAP_001.pdf